CLINICAL TRIAL: NCT05299047
Title: Fluoroscopic Anterior Approach Versus Ultrasound Guided Superior Hypogastric Plexus Neurolysis in Cancer Pelvic Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, assist. prof. of anesthesia and pain management, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R.22.01.1598
Record Dates: First submitted 2022-02-28; First posted 2022-03-28 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Pain Cancer
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group US-guided (Active Comparator): will receive superior hypogastric plexus neurolysis by the US-guided anterior approach
  Interventions: Other: Group US-guided
- - Group fluoroscopy-guided (Active Comparator): will receive superior hypogastric plexus neurolysis by the fluoroscopy-guided anterior approach
  Interventions: Other: Group fluoroscopy-guided

INTERVENTIONS:
Other: Group US-guided — An ultrasound system with a 5-2 MHz curved transducer will be used. The division of the abdominal aorta into the common iliac arteries was located using oblique sonography. Then, the transducer will image the body of the fifth lumbar vertebra, at which level bilateral common iliac vessels will be seen leaving a space in the midline. a 20 cm long, 22 gauge Chiba needle will be introduced into the hypogastrium, with out-of-plane technique to access the fifth lumbar vertebral body at its anterior-most point, so that injected drug spreads equally bilaterally along the anterior curvature of the fifth lumbar vertebral body.Suction was applied to the needle to confirm that it was not within a vessel and 10 ml of 50% ethanol will be injected for neurolysis.
  Arms: Group US-guided
Other: Group fluoroscopy-guided — The patient will be placed in the supine position. The L5-S1 inter-discal space was identified under fluoroscopy.After providing local cutaneous and subcutaneous anesthesia with 2% Lignocaine solution nearly 3-4 cm below the umbilicus, a 20 cm long, 22 gauges Chiba needle is advanced to the anterior portion of the 5th vertebral body under ongoing fluoroscopic guidance. Once bony resistance is reached, gently inject 2-5 ml contrast which typical reveals a characteristic triangular blob of contrast with no vascular opacification.Before injection the needle is aspirated to confirm there is no blood. A preliminary test dose of about 3 cc of 0.5% bupivacaine is then injected. If there is no change in heart rate or neurological status, rest of the 20 cc phenol 10% is injected slowly with intermittent aspiration.
  Arms: - Group fluoroscopy-guided

SUMMARY:
Cancer related pelvic pain can be debilitating and difficult to treat. Superior hypogastric plexus neurolysis (SHPN) is considered to be an option for adequately relieving pain, with fewer side effects and improving the quality of life

DETAILED DESCRIPTION:
The superior hypogastric plexus (SHP) is one of the paravertebral sympathetic ganglia, located in the lower border of the L5 vertebra and upper part of the sacrum in the retroperitoneal space. It is considered as a continuity of the celiac plexus and the lumbar sympathetic ganglia. It is related to the bifurcation of the aorta and the ureters. The SHP has a sympathetic connection (both efferent and afferent fibers) with splanchnic nerves and aortic plexus. It innervates the viscera of the pelvis, including the urinary bladder, ureters, sigmoid colon down to the anal canal, and upper vagina SHP blockade can be performed either by ultrasound (US), fluoroscopic, computed tomography (CT) and Magnetic resonance imaging (MRI) techniques and it is conducted through anterior (transabdominal) or posterior (lateral, paramedian, oblique, transdiscal, or transvaginal) approaches These different imaging modalities and approaches have been described for SHPN to make it easier, safer and more accurate and satisfied to the patients

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years old of both genders with cancer-related pelvic pain,
* poor pain control or severe side effects with opioid therapy,
* ≥ 4 on a numeric rating scale (NRS) of pain that ranged from 0 (no pain) to 10 (extreme pain).,
* American society of Anesthesiology Physical Status class I and II,
* positive diagnostic block day before the procedure by injecting a local anesthetic (0.25% bupivacaine 10 ml)
* Body mass index ˂ 30 were included in this study.

Exclusion Criteria:

* patient refusal,
* local or systemic sepsis,
* coagulopathy,
* unstable cardiovascular and respiratory diseases,
* previous neurological deficits,
* history of psychiatric disorders,
* history of drug abuse,
* distorted local anatomy,
* those who were allergic to the used medications were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
The symptom burden was evaluated using the Edmonton Symptom Assessment System (ESAS) | 0ne hour before block
  It includes the assessment of 10 symptoms experienced by cancer patients with the following 0-10 numeric rating scales: pain, fatigue, drowsiness, nausea, lack of appetite, depression, anxiety, shortness of breath, feeling of well-being, and insomnia.
The symptom burden was evaluated using the Edmonton Symptom Assessment System (ESAS) | 1 month from block
  It includes the assessment of 10 symptoms experienced by cancer patients with the following 0-10 numeric rating scales: pain, fatigue, drowsiness, nausea, lack of appetite, depression, anxiety, shortness of breath, feeling of well-being, and insomnia
The symptom burden was evaluated using the Edmonton Symptom Assessment System (ESAS) | 2 months from block
  It includes the assessment of 10 symptoms experienced by cancer patients with the following 0-10 numeric rating scales: pain, fatigue, drowsiness, nausea, lack of appetite, depression, anxiety, shortness of breath, feeling of well-being, and insomnia
The symptom burden was evaluated using the Edmonton Symptom Assessment System (ESAS) | 3 months from block
  It includes the assessment of 10 symptoms experienced by cancer patients with the following 0-10 numeric rating scales: pain, fatigue, drowsiness, nausea, lack of appetite, depression, anxiety, shortness of breath, feeling of well-being, and insomnia

SECONDARY OUTCOMES:
time of the procedures | intraoperative
  time of the procedure
daily analgesic requirements | 3 months from injection
  dose of opioid
patient satisfaction | 0ne month after block
  0 is very dissatisfied and 10 is very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Yahya Wahba, Al Mansurah, Egypt

REFERENCES:
- [Derived] Abdelghaffar NA, Farahat TE. Fluoroscopic anterior approach versus ultrasound guided superior hypogastric plexus neurolysis in cancer pelvic pain: a randomized controlled study. BMC Anesthesiol. 2022 Dec 27;22(1):403. doi: 10.1186/s12871-022-01948-3. PMID 36575390